CLINICAL TRIAL: NCT00499239
Title: Multi-center, Open-label, Dose-escalating Phase I/II Trial of GS-9219 Administered Once Every Three Weeks Intravenously to Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia, Non-Hodgkin's Lymphoma or Multiple Myeloma
Brief Title: A Trial of GS-9219 in Chronic Lymphocytic Leukemia (CLL), Non-Hodgkin's Lymphoma (NHL) or Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unacceptable safety profile
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-193-0101
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma
Keywords: Hematologic Malignancies; CLL; NHL; Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma; CLL and NHL; Multiple Myeloma; MM
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Hematologic Neoplasms | interventions — rabacfosadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GS-9219 (Experimental): Escalating doses of GS-9219 (5, 8, 11.5, 16, 22.5, 31.5, 44, and 61.5 mg/m^2) until determination of the maximum tolerated dose (MTD)
  Interventions: Drug: GS-9219

INTERVENTIONS:
Drug: GS-9219 — GS-9219 Injection is a clear, and colorless to slightly yellow aqueous solution containing 4 mg/mL of GS 9219.
  GS 9219 will be administered via IV infusion over 30 minutes in 100 mL of normal saline solution, every 21 days.

SUMMARY:
Multi-center, open-label, single-dose, dose-escalating Phase I/II study of GS 9219 in adult patients with relapsed or refractory CLL, NHL or MM. Patients will be enrolled into the study in sequential dose cohorts.

Patients will be administered a single IV infusion of GS 9219 on Day 1 of a 21 day cycle and may receive a total of six treatment cycles based on toxicities and response. Patients who demonstrate disease progression will be discontinued from the study. Patients who, at the completion of six treatment cycles, tolerate treatment and show evidence of disease control (response or stabilization) will be eligible to continue receiving treatment at the same dose.

DETAILED DESCRIPTION:
The primary objective of this study is as follows:

To assess the safety, toxicity, and maximum tolerated dose (MTD) of GS 9219 administered via IV administration once every three weeks (21 days) for six treatment cycles, i.e. for a total of 18 weeks, in patients with relapsed or refractory Chronic Lymphocytic Leukemia (CLL), Non-Hodgkin's Lymphoma (NHL) or Multiple Myeloma (MM).

The secondary objectives of this study are as follows:

To determine the pharmacokinetic parameters of GS 9219 for this regimen and patient population.

To assess the antitumor activity of GS 9219 based on Response Rate and Duration of Response. Progression-free Survival and Overall Survival will be assessed if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CLL, NHL or MM
* ECOG Performance Status of 0, 1, or 2
* Adequate organ function (protocol defined)
* ECG without evidence of clinically significant ventricular arrhythmias

Exclusion Criteria:

* AIDS-related lymphoma
* Subjects with NHL who present exclusively with non-measurable lesions
* Subjects with MM who have non-secretory and/or non-measurable disease
* Recent anticancer therapy (chemotherapy, radiotherapy, and/or biotherapy)within four weeks prior to starting treatment
* Evidence of pulmonary fibrosis
* Other concurrent malignancy
* Uncontrolled concurrent illness
* Receiving chronic, systemically administered steroids
* Known hypersensitivity to nucleoside analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Determination of MTD | All visits
  Toxicity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE). The MTD will be the highest dose level immediately below the dose level where two or more of three to six patients experience a dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Pharmacokinetics of GS-9219 and its metabolites | AAA) CLL/NHL: at Cycles 1, 3, and 6: MM: Cycles 1, 2, 3, 4, 5, and 6
  Pharmacokinetics (Cmax, Tmax, Clast, Tlast, λz, t1/2, AUClast, AUCinf, and %AUCexp) measured by blood sampling
Response rate | CLL/NHL: at Cycles 1, 3, and 6: MM: Cycles 1, 2, 3, 4, 5, and 6
  Response rate measured by:
  * CLL: National Cancer Institute Working Group (NCIWG) criteria
  * NHL - National Cancer Institute (NCI) criteria; Response Evaluation in
  * MM - International Myeloma Working Group (IMWG) criteria.
Duration of response | CLL/NHL: at Cycles 1, 3, and 6: MM: Cycles 1, 2, 3, 4, 5, and 6
  Duration of response measured by:
  * CLL: National Cancer Institute Working Group (NCIWG) criteria
  * NHL - National Cancer Institute (NCI) criteria; Response Evaluation in
  * MM - International Myeloma Working Group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hawkins, MD, Study Director — Gilead Sciences
Locations (20):
- United States (5):
  - UCSF, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada
  - MD Anderson Cancer Center, Houston, Texas
- Czechia (5):
  - Fakultni nemocnice Brno - Bohunice, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice, Prague
- Russia (10):
  - State Institution: Medical Radiological Research Center under the Russian Academy of Medical Sciences, Kaluga Region
  - State institution Main Military Clinical Hospital n.a.academician N.N. Burdenko under the Ministry of Defense of Russia, Moscow
  - State Institution Hematological Research Center under the Russian Academy of Medical Sciences, Moscow
  - Moscow State Medical Institution: Municipal Clinical Hospital n.a. S.P. Botkin, Moscow
  - Non-State Medical Institution Central Clinical Hospital #2 n.a. N.A. Semashko under OJSC "Russian Railways", Moscow
  - State Public Medical Institution of Novosibirsk Region: State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Federal State Institution: Research Institute of Hematology and Blood Transfusion under Federal Agency for High-Tech Medical Care, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University n.a. I.P. Pavlov under the Federal Agency for Healthcare and Social Development, Institute of Hematology and Transplantology n.a. R.M. Gorbacheva, Saint Petersburg
  - State Higher Educational Institution St. Petersburg State Medical University n.a. I.P. Pavlov under the Federal Agency for Healthcare and Social Development, Saint Petersburg
  - Federal State Institution Russian Research Center of Radiology and Surgical Technologies under the Federal Agency for High-Tech Medical Care, Saint Petersburg